CLINICAL TRIAL: NCT05036343
Title: Smart Insulin Pens: A Randomized, Crossover Prospective Interventional Pilot Study Assessing the Effect on Glycemic Control and Diabetes Related Burdens
Brief Title: A Study to Assess the Effect of Smart Insulin Pens on Glycemic Control and Diabetes-related Burdens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Ana L. Creo, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 21-004938
Record Dates: First submitted 2021-09-02; First posted 2021-09-05 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Type 1 Diabetes
Keywords: Adolescents; Young Adults; Continuous Glucose monitoring (CGM)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- InPen® and CGM, then standard of care and CGM (Experimental): Adolescents and young adults (13-21 years) identified with having type 1 diabetes and currently receiving insulin injections with a continuous glucose monitor (CGM) will use the InPen® and CGM for the first 90 days then switch to standard of care with traditional insulin injections and CGM for 90 days.
  Interventions: Device: InPen®
- Standard of care and CGM, then InPen® and CGM (Experimental): Adolescents and young adults (13-21 years) identified with having type 1 diabetes and currently receiving insulin injections with a continuous glucose monitor (CGM) will receive standard of care with traditional insulin injections and CGM for first 90 days then switch to the InPen® and CGM for 90 days.
  Interventions: Device: InPen®

INTERVENTIONS:
Device: InPen® — A smartpen that has been FDA approved for children with diabetes age seven years and older that uses an app on a smartphone to help calculate insulin doses using the amount of carbohydrates that will be consumed at a meal along with what the current blood sugar reading is, to give a correction dose as well. The InPen app also serves as a log book to record insulin doses given, blood sugar at the time of a meal, and amount of carbohydrate eaten.

SUMMARY:
The purpose of this study is to see if the use of the InPen® for teens and young adults up to age 21 years with type 1 diabetes helps to decrease burden and improve glycemic control.

DETAILED DESCRIPTION:
Investigators will perform a randomized, cross-over prospective interventional study. Half of the participants will be randomized to the InPen® and the other half will continue with their conventional insulin injection protocol. After 90 days, participants will switch to the second arm. Randomization will occur via block randomization. Teaching to use the InPen® will be done by Sarah Jackson, DO with supervision by Ana Creo, MD, which can be done by a telemedicine visit if it does not align with clinic visit. You will be followed for three months with hemoglobin A1c at the beginning and the end of the study. Data from the (Continuous Glucose Monitor (CGM) and InPen® will be analyzed including time in glucose goal range (70-180 mg/dL), glucose standard deviation, percentage of time that is spent high (>180-250 mg/dL), very high(> 250 mg/dL), low(54-70 mg/dL) and very low(<54 mg/dL), along with total daily insulin dose. Data on missed insulin doses will be assessed via data from the InPen®. You will be randomized to traditional injections we will ask them to record missed insulin doses weekly. You should still adjust insulin doses at home, like they do at baseline. If insulin adjustments are made while in one arm of the study they should still continue that dosing when they cross over. Investigators will also assess quality of life and fatigue related to technology with surveys prior to start of the study and at the end. Specifically, investigators will assess diabetes distress, transition readiness, and parental experience of childhood illness scales. Investigators will also utilize the insulin delivery satisfaction survey to assess how you view your current regimen and then how you view the effects of the InPen in managing your type 1 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Individuals between the ages of 13 and 21 years.
* Patients with Type 1 diabetes for at least 6 months
* Defined as either a c peptide <1 , one or more positive diabetes autoantibodies, or a clinical diagnosis with age of onset prior to puberty
* Patients who currently receive insulin injections with a CGM.
* English speaking.
* Have access to a smart phone. on an insulin to carbohydrate ratio

Exclusion Criteria:

* Individuals less than 13
* Non-English speaking.
* No access to a smart phone.
* Intellectual disability that would impact their ability to utilize the technology
* Known pregnant women taking chronic steroids (equivalent equal to or greater then 5mg of prednisone daily)

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 13 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2022-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Creo, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials

RESULTS

PARTICIPANT FLOW:
Groups:
- InPen® and CGM, Then Standard of Care and CGM: Adolescents and young adults (13-21 years) identified with having type 1 diabetes and currently receiving insulin injections with a continuous glucose monitor (CGM) used the InPen® and CGM for the first 90 days then switched to standard of care with traditional insulin injections and CGM for 90 days.
  InPen®: A smartpen that has been FDA approved for children with diabetes age seven years and older that uses an app on a smartphone to help calculate insulin doses using the amount of carbohydrates that will be consumed at a meal along with what the current blood sugar reading is, to give a correction dose as well. The InPen app also serves as a log book to record insulin doses given, blood sugar at the time of a meal, and amount of carbohydrate eaten.
- Standard of Care and CGM, Then InPen® and CGM: Adolescents and young adults (13-21 years) identified with having type 1 diabetes and currently receiving insulin injections with a continuous glucose monitor (CGM) received standard of care with traditional insulin injections and CMG for first 90 days then switched to the InPen® and CMG for 90 days.
  InPen®: A smartpen that has been FDA approved for children with diabetes age seven years and older that uses an app on a smartphone to help calculate insulin doses using the amount of carbohydrates that will be consumed at a meal along with what the current blood sugar reading is, to give a correction dose as well. The InPen app also serves as a log book to record insulin doses given, blood sugar at the time of a meal, and amount of carbohydrate eaten.
Period: First Intervention (90 Days)
Arm/Group | InPen® and CGM, Then Standard of Care and CGM | Standard of Care and CGM, Then InPen® and CGM
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0
Period: Second Intervention (90 Days)
Arm/Group | InPen® and CGM, Then Standard of Care and CGM | Standard of Care and CGM, Then InPen® and CGM
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- InPen® and CGM, Then Standard of Care and CGM: Adolescents and young adults (13-21 years) identified with having type 1 diabetes and currently receiving insulin injections with a continuous glucose monitor (CGM) used the InPen® and CMG for the first 90 days then switched to standard of care with traditional insulin injections and CMG for 90 days.
  InPen®: A smartpen that has been FDA approved for children with diabetes age seven years and older that uses an app on a smartphone to help calculate insulin doses using the amount of carbohydrates that will be consumed at a meal along with what the current blood sugar reading is, to give a correction dose as well. The InPen app also serves as a log book to record insulin doses given, blood sugar at the time of a meal, and amount of carbohydrate eaten.
- Total: Total of all reporting groups
Arm/Group | InPen® and CGM, Then Standard of Care and CGM | Standard of Care and CGM, Then InPen® and CGM | Total
Number analyzed (Participants) | 5 | 8 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.0 (1.22) | 15.9 (1.89) | 15.9 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 5 | 6 | 11
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 8 | 13

OUTCOME MEASURES:

1. Primary Outcome: Glucose Time in Range
Description: The percentage of time that glucose readings are in goal range (70-180 mg/dL)
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: percentage of time in range
Groups:
- InPen® and Continues Glucose Monitoring (CGM): Subjects who received InPen® and CGM in either the first or last 90 days of the study
- Standard of Care and Continues Glucose Monitoring (CGM): Subjects who received standard of care and CGM in either the first or last 90 days of the study
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 13
percentage of time in range | 46 (22) | 49 (20)

2. Primary Outcome: InPen® Missed Insulin Injections
Description: Number of missed insulin injections after 30 and 90 days of InPen and CGM
Time Frame: 30 and 90 days
Population: Only InPen & CGM subjects data were collected and analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: missed insulin injections
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 0
missed insulin injections
  30 days | 51.2 (26.3) |
  90 days | 212.6 (76.1) |

3. Primary Outcome: Change in Hemoglobin A1c
Description: Hemoglobin is a protein within red blood cells. As glucose enters the bloodstream, it binds to hemoglobin, or glycates. The more glucose that enters the bloodstream, the higher the amount of glycated hemoglobin. An A1C level below 5.7 percent is considered normal. Unit of measure = percent of glycated hemoglobin
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: percent of glycated hemoglobin
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 13
percent of glycated hemoglobin | -0.1 (0.6) | -0.3 (0.7)

4. Primary Outcome: Glucose
Description: Mean glucose levels at 6 months. Sugar in the form of glucose in the blood. The concentration of glucose in the blood. A healthy normal range is 70 to 99 mg/dL
Time Frame: 3 months
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 13
mg/dL | 198 [178 to 212] | 180 [167 to 213]

5. Secondary Outcome: Change in Diabetes Distress Scale Score
Description: Measured using the Diabetes Distress Scale (DDS) which identifies 17 potential problem areas that people with diabetes may experience and asked subjects to rate their perceived degree of distressed during the past month; using a scale of 1 = "Not a problem at all", 6 = "A very serious problem." Total scores range from 17-102, lower scores indicating less distress and higher scores indicating more distress
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 13
score on a scale | -0.038 (0.231) | 0.075 (0.283)

6. Secondary Outcome: Change in Transition Readiness
Description: Mean change in transition readiness as measured by using the Transition Readiness Assessment Questionnaire (TRAQ). A 20-item questionnaire assessing the skill levels that are important for transition to adult health care; using a scale of 1 = "No, I do not know how", 5 = "Yes, I always do this when I need to." Total scores range from 20 - 100, lower scores indicating lower readiness and higher scores indicating greater readiness.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 13
score on a scale | 0.149 (0.785) | -0.029 (0.739)

7. Secondary Outcome: Change in Self-Efficacy for Managing Chronic Conditions - Managing Medications and Treatment Score
Description: Measured using the Self-Efficacy for Managing Chronic Conditions - Managing Medications and Treatment questionnaire. A 14-item questionnaire rating the confidence level for managing chronic conditions, medications and treatment; using a scale of 1 = "I am not at all confident", 5 = "I am very confident." Total scores range from 14-70, lower scores indicating lower confidence and higher scores indicating higher confidence.
Time Frame: Baseline, 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
Number analyzed (Participants) | 13 | 13
score on a scale | 0.058 (0.464) | 0.074 (0.514)

ADVERSE EVENTS:
Time Frame: Adverse Events were assessed for all subjects during first treatment period (90 days) and second treatment period (90 days) for a total of approximately 6 months.
Arm/Group | InPen® and Continues Glucose Monitoring (CGM) | Standard of Care and Continues Glucose Monitoring (CGM)
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/13
Other Adverse Events (participants affected / at risk) | 0/13 | 0/13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT05036343/Prot_SAP_000.pdf